CLINICAL TRIAL: NCT06556251
Title: Evaluating the Effectiveness of a Digital Platform in the Engagement and Prognosis of Patients in the Early Intervention Programme in Psychosis
Brief Title: Effectiveness of a Digital Platform in Engagement and Prognosis of Patients in an Early Intervention Pychosis Programme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PIC_37_23
Record Dates: First submitted 2024-07-02; First posted 2024-08-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-12

CONDITIONS: Device Adherence
Keywords: platform; technologies; young people; early psychosis; adherence
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This study will be a randomised, prospective and single-centre clinical trial in which one group (EG) will have access to the PIPPEP platform in addition TAU, while the other group (CG) will receive TAU without using the platform.
  The study will be carried out in all 9 community mental health centres of the Sanitary Parc Sant Joan de Déu. Patients will be randomly assigned to the EG or CG using a list of random numbers. The evaluation will be based on variables of the clinical history of the patients in both conditions (EG and CG) at the beginning of the study, after 6 months and after 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental group (EG) will have access to the PIPPEP platform in addition to treatment in the Early Psychosis Programme.
  Interventions: Device: PIPPEP App
- Treatment as Usual (Active Comparator): The control group (CG) will receive treatment as usual (TAU) without using the platform.
  Interventions: Device: PIPPEP App

INTERVENTIONS:
Device: PIPPEP App — Digital platform with psichoeducative content in infographics, animated and testimonial videos about:
  * psychotic and comorbid symptoms, substance use, available treatments, healthy lifestyle habits, social and health emergency resources and outpatient clinics for young people.
  * Regular self-completed questionnaires to measure alarm symptoms, side effects of pharmacological treatment, emotional state, and treatment adherence. There will be a feedback for patients in the form of graphs of the evolution of the different types of questionnaires.
  * A bidirectional messaging service with the professional reference team, allowing better accessibility in non-urgent cases.
  * A gamification system to encourage use of the application, which includes points, rewards, a leaderboard and mini-games.
  * A folder where patients can keep documents they find useful (personal reports, relapse prevention plan, crisis plan).

SUMMARY:
This is a randomised, prospective, controlled trial in which one group (experimental group; GE) receives access to the PIPPEP (Intervention Programme for Early Psychosis) platform in addition to the treatment as usual (TAU) in PIPPEP, while the other group (control group; GC) receives only TAU in PIPPEP.

Main objective:

- To assess whether the use of the PIPPEP platform improves psychosocial and pharmacological treatment adherence in mental health programmes.

Secondary objectives:

* To assess the cost-effectiveness of the PIPPEP app.
* Evaluation of the dissemination of the platform.
* To assess the clinical and functional outcomes of patients using the PIPPEP platform in terms of 1) positive symptoms, 2) side effects of antipsychotic medication, 3) perceived social self-stigma, 4) risk assessment, 5) comorbid symptoms and 6) social functioning

The participants are 1) between 18 and 40 years of age, who are being treated in one of the PIPPEP programmes for early intervention in psychosis at Sanitary Parc Sant Joan de Déu and who meet the inclusion criteria "extremely high risk of psychosis", "critical phase or "first psychotic episode" and 2) agree to participate in the study and sign the informed consent form.

DETAILED DESCRIPTION:
Background:

Mental disorders are the most common cause of disability in young people, with the disconnect with mental health in adolescents being as high as 50% in some cases. Much research has been conducted on psychotic disorders in recent decades, particularly on their early clinical manifestations. This has led to the establishment of numerous psychosis detection and early intervention programmes around the world to initiate treatment as early as possible.

This situation emphasises the need to change the model of mental health care and focus on the adolescent population in particular with preventive, diagnostic and therapeutic interventions. To improve patient engagement, the importance of a good therapeutic alliance, patient voluntarism, a collaborative approach and clear and continuous communication between patients and professionals was emphasised.

Online and mobile interventions have been shown to be acceptable and effective in improving individuals' self-care practises across a wide range of healthcare settings. They have enabled the implementation of evidence-based interventions to promote healthy behaviours (smoking cessation, physical activity, anxiety, depression...) and reduce barriers to accessing mental health services, and have also been shown to be feasible, acceptable and effective for a wide range of mental health conditions. Ease of use, accessibility and potentially reduced stigmatisation are cited as benefits. They also have the potential to reduce healthcare costs and offer options to aid diagnosis, facilitate real-time assessment and monitoring of symptoms, and provide innovative treatments for a variety of conditions. Adherence rates for these interventions are high, ranging from 60-100% (average 83%). A recent Canadian study conducted with a sample of young people treated in an early intervention team concluded that the use of the internet and various technological devices by young people with a first episode of psychosis is similar to that of young people in the general population of the same age.

Procedure:

This study will be a randomised, prospective and single-centre clinical trial in which one group (EG) will have access to the PIPPEP platform in addition to treatment in the PIPPEP, while the other group (CG) will receiveTAU without using the platform.

A second part of the study will consist of a quasi-experimental longitudinal study of a single group (EG) in which the data from the questionnaires submitted via the platform will be analysed. The data from the questionnaires will be transferred to and stored in each participant's medical record, with all the security measures that apply to all patient data.

These questionnaires will appear in a notification format on the participant's device and will be completed at the beginning of the study, after 6 months and after 12 months, with the exception of the anxiety and depression questionnaire, which will be completed weekly.

Interventions:

The PIPPEP is a care programme that includes patients with a first psychotic episode (FEP), with a UHR or within the first 5 years of illness development (critical period). It is a multidisciplinary intervention involving psychiatric, nursing, social work and psychological visits using evidence-based psychotherapy (cognitive-behavioural). The maximum duration of the intervention is 5 years.

Patients belonging to the EG will additionally have access to the PIPPEP platform, while patients assigned to the CG will continue to receive TAU. The platform will have the basic functionalities already present in the PIPPEP application (requesting reports, visits or tests) and will also include the following content:

* Specific information about psychotic and comorbid symptoms, substance use, available treatments, healthy lifestyle habits, knowledge of emergency social and health resources, and outpatient clinics for youth. The psychoeducational content will include links that redirect to the SOM 360 (Mental Health webpage) (specifically the psychosis website) for more in-depth information.
* Additional questionnaires that will be self-completed at regular intervals to allow the clinical team to monitor symptoms, emotional state, side effects, etc. The information obtained through these questionnaires is transmitted directly and stored in each patient's medical history, with all the associated security measures.
* A bi-directional messaging service with the referral team to allow better accessibility for non-urgent aspects.
* A reward system to encourage use of the application with points, rewards and mini-games.
* A folder where patients can keep documents they find useful, such as the relapse prevention plan and the crisis plan.

In addition, during the personalised follow-up sessions that are part of the TAU, patients assigned to the EG will receive support in using the application from the PIPPEP therapists.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 40 years
* Fulfil the criteria for one of the three groups (First Psychotic Episodes, Critical Period or Ultra High Risk of Psychosis; UHR)
* To undergo community-based treatment as part of one of our facility's early intervention programmes for psychosis
* Have signed the informed consent form for the study.

Exclusion criteria:

* No mobile phone/laptop/tablet to use the platform.
* Lack of skills and/or knowledge to use the platform.
* Not have knowledge of the Catalan or Spanish language.
* Have a diagnosed mental disability (premorbid Intelligence Quotient <70).
* Have had a medical condition that better explains the psychotic symptoms.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to psychosocial treatment. | Baseline, 6 months follow-up, 12 months follow-up
  Attendance at follow-up appointments with the therapeutic team. Lack of engagement or lack of adherence will be assumed if the patient remains uninterrupted for a period of at least one month despite the need for treatment:
  1. does not turn up for scheduled visits and does not report in.
  2. cannot be reached by telephone.
  3. actively refuses contact with professionals and/or treatment.
  If one of the above conditions is met, the person's last contact is considered the date of drop-out.

SECONDARY OUTCOMES:
Direct costs use services | Baseline, 6 months follow-up, 12 months follow-up
  Direct costs related to the use of services (e.g. scheduled primary care visits, urgent General Practitioner visits,tests (TAC, Magnetic Resonance, Analytical).
Penetration of the platform | Baseline, 6 months follow-up, 12 months follow-up
  Penetration of the platform (e.g. number of accesses to the platform, number of consultations with professionals).
Indirect costs | Baseline, 6 months follow-up, 12 months follow-up
  Indirect costs (e.g. temporary inability to work, permanent disabilities, premature mortality (completed suicide, accident, other medical causes).
Scale of the Impact of Perceived Symptoms in Schizophrenia | Baseline, 6 months follow-up, 12 months follow-up
  This is a self-administered scale that measures psychotic symptoms and the impact of symptoms on the patient's daily life.
Medication Adherence Scale-8 items | Baseline, 6 months follow-up, 12 months follow-up
  It is a 8 items is a structured, self-administered measure of medication adherence behaviour. It consists of 8 items and asks the person to answer yes or no to questions about medication adherence. Total scores are categorized as low (MMAS-8 score <6), medium (MMAS-8 score 6 to <8), and high (MMAS-8 score 8). Lower scores indicate worse adherence.
Scale for side effects of medication (UKU) | Baseline, 6 months follow-up, 12 months follow-up
  This scale evaluates psychological, neurological, autonomic and other side effects of the medication. At the end there is a general assessment of the impairment that these effects may have on the patient's daily activities.It comprises ratings (0-4) of 48 single items, the higher the score, the greater the presence and severity of side effects.
The Beck Cognitive Insight Scale for Schizophrenia (BCIS) | Baseline, 6 months follow-up, 12 months follow-up
  It is a self-administered scale that measures cognitive insight capacity, i.e., self-reflection as a metacognitive mechanism for analysing the symptoms of the illness that allows for continuous re-evaluation of inappropriate interpretations. A composite index, Cognitive Insight, is calculated as Reflectiveness minus Certainty (CI=R-C). The response format includes four Likert-type options: Never Agree (0), Somewhat Agree (1), Quite Agree (2) and Totally Agree (3), with a total score between 0 and 45. Higher scores on self-reflection and the composite index indicate greater cognitive insight, while lower scores on self-confidence indicate better cognitive insight.
Questionnaire on the consumption of toxic substances | Baseline, 6 months follow-up, 12 months follow-up
  Ad hoc checklist asking to indicate whether the person has consumed any of the following substances in the last 3 months: Caffeine or theine, tobacco, alcohol, cannabis, cocaine, amphetamines, opiates, hallucinogens, designer drugs, stimulants, benzodiazepines, inhalants or other drugs. The participant will be also asked to indicate the quantity and frequency of use.
Questionnaire on anxiety and depression | Baseline, 6 months follow-up, 12 months follow-up
  It consists of two ad hoc questions in which the person is asked a) to what extent they have felt nervous and/or stressed in the last week and b) to what extent they have felt sad and/or depressed. The person must answer on a scale from 0 to 5: "never", "almost never", "occasionally", "often" or "very often". The higher the score, the greater the presence and severity of the side effects
Scale for self-perception of social stigmatisation (SSQ) | Baseline, 6 months follow-up, 12 months follow-up
  This is a self-administered scale with a number of statements relating to the respondent's views on mental illness and their own experiences. It is required that the level is chosen according to the statements presented, on a scale of 1 to 7 (1 = Strongly agree, 2 = moderately agree, 3 = slightly agree, 4 = neither agree nor disagree, 5 = slightly disagree, 6 = moderately disagree, and 7 = strongly disagree). Higher scores indicate lower self-stigma.
Quality of life. Quality of Life Index (QLI-sp) | Baseline, 6 months follow-up, 12 months follow-up
  This is a 10-item questionnaire covering the following dimensions: psychological well-being, physical well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, emotional and social support, community support and services, self-actualisation or personal fulfilment, spiritual satisfaction and global quality of life assessment. Each item is rated by the respondent according to their personal and cultural view of this concept on a Likert scale from 0 to 10 points. The higher the score, the higher the respondent's quality of life.
Global Assessment of Functioning (GAF) scale | Baseline, 6 months follow-up, 12 months follow-up
  It is an heteroadministered scale that assesses the patient's functioning (including psychological, social and occupational activities) over the last 12 months on a scale between 0 and 100. Higher scores indicate higer level of functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Lal S, Malla A. Service Engagement in First-Episode Psychosis: Current Issues and Future Directions. Can J Psychiatry. 2015 Aug;60(8):341-5. doi: 10.1177/070674371506000802. PMID 26454555
- [Background] Lloyd-Evans B, Sweeney A, Hinton M, Morant N, Pilling S, Leibowitz J, Killaspy H, Tanskanen S, Totman J, Armstrong J, Johnson S. Evaluation of a community awareness programme to reduce delays in referrals to early intervention services and enhance early detection of psychosis. BMC Psychiatry. 2015 May 2;15:98. doi: 10.1186/s12888-015-0485-y. PMID 25934413
- [Background] Marshall M, Rathbone J. Early intervention for psychosis. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD004718. doi: 10.1002/14651858.CD004718.pub3. PMID 21678345
- [Background] Leclerc E, Noto C, Bressan RA, Brietzke E. Determinants of adherence to treatment in first-episode psychosis: a comprehensive review. Braz J Psychiatry. 2015 Apr-Jun;37(2):168-76. doi: 10.1590/1516-4446-2014-1539. Epub 2015 May 1. PMID 25946398
- [Background] Bonsack C, Pfister T, Conus P. [Linkage to care after first hospitalisation for psychosis]. Encephale. 2006 Oct;32(5 Pt 1):679-85. doi: 10.1016/s0013-7006(06)76219-4. French. PMID 17099591
- [Background] Schimmelmann BG, Conus P, Schacht M, McGORRY P, Lambert M. Predictors of service disengagement in first-admitted adolescents with psychosis. J Am Acad Child Adolesc Psychiatry. 2006 Aug;45(8):990-999. doi: 10.1097/01.chi.0000223015.29530.65. PMID 16865042
- [Background] Berry D, Blair C, Willoughby M, Garrett-Peters P, Vernon-Feagans L, Mills-Koonce WR; Family Life Project Key Investigators. Household Chaos and Children's Cognitive and Socio-Emotional Development in Early Childhood: Does Childcare Play a Buffering Role? Early Child Res Q. 2016 1st Quarter;34:115-127. doi: 10.1016/j.ecresq.2015.09.003. Epub 2015 Oct 31. PMID 29720785
- [Background] Arean PA, Hoa Ly K, Andersson G. Mobile technology for mental health assessment. Dialogues Clin Neurosci. 2016 Jun;18(2):163-9. doi: 10.31887/DCNS.2016.18.2/parean. PMID 27489456
- [Background] Torous J, Roux S. Patient-Driven Innovation for Mobile Mental Health Technology: Case Report of Symptom Tracking in Schizophrenia. JMIR Ment Health. 2017 Jul 6;4(3):e27. doi: 10.2196/mental.7911. PMID 28684386
- [Background] Gay C, Chabaud A, Guilley E, Coudeyre E. Educating patients about the benefits of physical activity and exercise for their hip and knee osteoarthritis. Systematic literature review. Ann Phys Rehabil Med. 2016 Jun;59(3):174-183. doi: 10.1016/j.rehab.2016.02.005. Epub 2016 Apr 1. PMID 27053003
- [Background] Abdel-Baki A, Lal S, D-Charron O, Stip E, Kara N. Understanding access and use of technology among youth with first-episode psychosis to inform the development of technology-enabled therapeutic interventions. Early Interv Psychiatry. 2017 Feb;11(1):72-76. doi: 10.1111/eip.12250. Epub 2015 May 22. PMID 26011657
- [Background] Killikelly C, He Z, Reeder C, Wykes T. Improving Adherence to Web-Based and Mobile Technologies for People With Psychosis: Systematic Review of New Potential Predictors of Adherence. JMIR Mhealth Uhealth. 2017 Jul 20;5(7):e94. doi: 10.2196/mhealth.7088. PMID 28729235